CLINICAL TRIAL: NCT02461797
Title: Evaluation of Nasal Mucosal Permeability in Controls and House Dust Mite Allergic Rhinitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: biopsystudy
Record Dates: First submitted 2015-04-27; First posted 2015-06-03 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-04

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- healthy controls (Other): biopsy of nasal mucosa healthy controls
  Interventions: Other: healthy controls
- AR patients with use of nasal corticoid spray (Other): biopsy of nasal mucosa allergic rhinitis to house dust mite with nasal corticosteroid spray
  Interventions: Other: AR patients with use of nasal corticoid spray
- AR patients without medication (Other): biopsy of nasal mucosa allergic rhinitis to house dust mite without any use of medication for symptom control
  Interventions: Other: AR patients without medication

INTERVENTIONS:
Other: healthy controls — biopsy of nasal mucosa for healthy controls
  Arms: healthy controls
Other: AR patients without medication — biopsy of nasal mucosa for allergic rhinitis patients without allergy medication
  Arms: AR patients without medication
Other: AR patients with use of nasal corticoid spray — biopsy of nasal mucosa for allergic rhinitis patients with use of nasal corticoid spray
  Arms: AR patients with use of nasal corticoid spray

SUMMARY:
Recently, a critical role in the development of allergic rhinitis (AR) has been attributed to the nasal epithelium. The airway epithelium forms a physical barrier, protecting the nasal mucosa and underlying organs from damage from contact with exogenous particles. The nasal epithelial barrier is primarily determined by the integrity of the airway epithelium, in which epithelial cells are connected to each other by complex network structures like tight junctions (TJs), ultimately sealing off the paracellular space. TJs consist of different transmembrane proteins including occludin, tricellulin, the claudin family, and junctional adhesion molecules. TJ form intercellular homodimers/heterodimers between neighboring cells. Scaffold adaptor proteins like cingulin and the zonula occludens family connect the transmembrane proteins to the actin cytoskeleton.

Disturbed TJ function can facilitate the entrance of foreign pathogens and antigens into the submucosal layer, giving raise to allergic sensitization via increased access of allergens to the dendritic cells and/or inducing persistent inflammation via activation of mast cells and other inflammatory cells residing in the upper airways. Chronic disorders like allergic asthma, inflammatory bowel disease and atopic dermatitis have been linked to defective or altered TJ function. Recently, an impaired epithelial barrier function was found in patients with chronic rhinosinusitis with nasal polyps (CRSwNP), suggesting changes in TJ arrangement in the nasal cavity. CRSwNP presents a similar inflammation of the sinonasal cavities as found in AR patients, i.e. a Th2 cytokine driven inflammation with tissue eosinophilia. Nevertheless, the role of TJs and its regulation has not been investigated in AR.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an ARIA-based diagnosis of persistent moderate/severe AR (≥ 2 nasal symptoms suggestive of allergic rhinitis and positive skin prick tests to HDM (HAL Allergy, Leiden, The Netherlands), and with VAS score for total nasal symptoms of more than 5
2. Age > 18 and < 60 years.
3. Possibility to give reliable information and written informed consent
4. For AR group with nasal corticosteroid spray: Patients that use nasal corticosteroid spray for at least three weeks prior to the study, with a minimum application of two puffs per nostril once a day.

Exclusion Criteria:

1. No common cold in the last 4 weeks
2. Patients on prolonged use of decongestive nose sprays, suffering from so-called rhinitis medicamentosa
3. A. For healthy controls and AR without use of nasal spray: Patients using other nasal or oral medication affecting nasal function, like nasal corticosteroids, anticholinergics, cromoglycates, leukotriene antagonists, ACE inhibitors less than 4 weeks before start of the study.

   B. For AR group with use of nasal corticosteroid spray: Patients using other nasal or oral medication affecting nasal function, like anticholinergics, cromoglycates, leukotriene antagonists, ACE inhibitors less than 4 weeks before start of the study.
4. Nasal endoscopic evidence of rhinosinusitis w/wo NP or structural abnormalities such as clinically relevant septal deviation (septum reaching concha inferior or lateral nasal wall) or septal perforation
5. Patients on immunotherapy (IT) for house dust mite (HDM) or with history of IT for HDM
6. Patient with a psychiatric, addictive, or any disorder of which the investigators feel that this may compromise the ability to give truly informed consent for participation in this study or provide reliable information on the questionnaire
7. Patients being enrolled in other clinical trials
8. Pregnancy or breastfeeding
9. Malignancies or severe comorbidity
10. Contra-indication for local anesthesia with cocaine 5%
11. Smoking
12. Use of anticoagulation medication

Healthy controls will meet the same exclusion criteria, with additional inclusion criteria:

1. Absence of nasal symptoms
2. Negative history of respiratory allergy
3. Negative skin prick test (SPT) results

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
change in Transepithelial electrical resistance (TEER) | every 30 min over 2 hours
  Nasal biopsies will be mounted in modified 3 ml Ussing chambers. Experiments will be performed in open-circuit conditions. Transepithelial electrical resistance (TEER) will be calculated from the voltage deflections induced by bipolar constant-current pulses of 16 mA every 60 s with duration of 200 ms and will be recorded every 30 min over 2 h. The average of all time points of the 2 biopsy samples/patient will be used and will be presented as Ωxcm².
change in mucosal permeability | every 30 min over 2 h
  The paracellular probe, fluorescently labelled dextran 4 kDa (FD4) (2 mg/ml) will be used to determine the mucosal permeability. FD4 will be added to the mucosal compartment and serosal samples will be collected every 30 min over 2 h. The fluorescence level will be measured using a fluorescence reader. The average of time points 60, 90 and 120 min of the 2 biopsy samples/patient will be used to express mucosal permeability.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hellings, MD PhD, Principal Investigator — UZ Leuven
Locations (1):
- ORL, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Steelant B, Farre R, Wawrzyniak P, Belmans J, Dekimpe E, Vanheel H, Van Gerven L, Kortekaas Krohn I, Bullens DMA, Ceuppens JL, Akdis CA, Boeckxstaens G, Seys SF, Hellings PW. Impaired barrier function in patients with house dust mite-induced allergic rhinitis is accompanied by decreased occludin and zonula occludens-1 expression. J Allergy Clin Immunol. 2016 Apr;137(4):1043-1053.e5. doi: 10.1016/j.jaci.2015.10.050. Epub 2016 Feb 2. PMID 26846377